CLINICAL TRIAL: NCT03690895
Title: Long-term Outcome of AIDS-related Primary Central Nervous System Lymphoma Treated With High Dose Methotrexate and Combined Antiretroviral Therapy
Acronym: LCPVIH
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_2015_2_AMR
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Central Nervous System Lymphoma; AIDS Related Lymphoma
MeSH Terms: conditions — Lymphoma, AIDS-Related

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases
  Interventions: Other: Retrospective survival analysis

INTERVENTIONS:
Other: Retrospective survival analysis — Kaplan-Meier model

SUMMARY:
This study aims at describing survival rates over time (Kaplan-Meier estimator) in patients suffering from AIDS-related primary central nervous system lymphoma who were diagnosed from 1996 to 2014 and treated with infusions of high-dose methotrexate and combined antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* AIDS-related primary central nervous system lymphoma
* treated with at least one infusion of methotrexate and combine antiretroviral therapy

Exclusion Criteria:

* prior non-Hodgkin lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for AIDS-related primary central nervous system lymphoma in Fondation Rothschild (Paris, France) between january1996 and december 2014
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Median duration of survival after diagnosis of lymphoma (years) | At the time of systematic files review (jan 2014) - average follow-up 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France

IPD SHARING:
Plan to Share IPD: No